CLINICAL TRIAL: NCT02512107
Title: The Effect of Juice Plus+ on the Microbiome, Intestinal Permeability and Inflammatory Status of Psychologically Stressed Individuals With High Body Mass Indices
Brief Title: Impact of JuicePlus+ on the Health Status of an Overweight Stressed Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 560061
Record Dates: First submitted 2015-07-01; First posted 2015-07-30 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Juice Plus+ (Active Comparator): Subject will be taking supplement.
  Interventions: Dietary Supplement: Juice Plus+
- Placebo (Placebo Comparator): Subjects will be taking the placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Juice Plus+ — Dried fruit and vegetable juice capsule.
  Arms: Juice Plus+
Other: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if a dried fruit and vegetable supplement (Juice Plus+) can alter the gut microbiome and improve gut permeability and inflammatory levels in an obese, stressed population.

The microbiome and its component genes are long known as critical determinants of the nutritional value of the food we eat. Recently, it has become clear that the composition of this microbiome and its metabolites influences the host immune system, thereby altering host physiology. Both obesity and chronic stress have been shown to have an altered gut microbiome; both these conditions also lead to increased systemic inflammatory molecules that can lead to an increased risk for type 2 diabetes and other diseases caused by chronic inflammation.

Juice Plus+ consumed by an overweight population combined with an eight week exercise regime showed decreased markers of protein/lipid oxidation (ox-LDL), total lipid oxidation (TOS) and lowered systemic concentrations of the inflammatory cytokine, TNF-α. As systemic cytokines are altered by the composition of the gut microbiome, this study proposes to determine if this decrease in inflammation by Juice Plus+ is due to a change in the species composition and metabolism of the microbiome. This question is particularly relevant for populations with high inflammatory loads resulting from excess weight in addition to increased psychological stress.

The investigators propose to determine 1) how Juice Plus+ consumption alters the microbiome species composition and metabolism, 2) if there is an alteration in intestinal permeability with the consumption of Juice Plus+ and 3) do these alterations coincide with lower systemic markers of inflammation and oxidative stress among individuals who are psychologically stressed and overweight. The investigators will use a randomized, placebo-controlled design with a cohort of overweight, female, critical care health care professionals. Subjects will receive the supplements or placebo for sixteen weeks. At the end of 16 weeks, the cohort receiving the supplement will be randomized to also receive a meal replacement component or follow their normal diet for an additional 4 weeks. Stool and a fasting blood sample will be collected at the beginning of the study (baseline) and 8, 16 and 20 weeks later. At each time point, subjects will also consume a cocktail of glucose, mannitol and lactulose and a second blood draw performed to look at absorption of these molecules.

DETAILED DESCRIPTION:
An anticipated eighty critical care, female health care professionals will be recruited. This population has been shown to have a high occupational stress load and have increased risk for post-traumatic stress disorder (PTSD). The subjects will be premenopausal, overweight/obese (Body Mass Index -BMI : 25 - 40 kg/m2) and between the ages of 25-50 years.

Exclusion criteria include smoking of any sort, smokeless tobacco use, chronic or excessive alcohol consumption (>1 drink per day), pregnancy or lactation, recent surgery or illness, diabetes, heart disease, use of antibiotics or medications (other than medication deemed not to impact outcome measures in this protocol-medication use will be reviewed on a case by case basis by the principal investigator).

Health history, medication and dietary supplement questionnaires will be completed by all subjects to determine eligibility. A health and perceived stress questionnaire will also be completed at each sampling period. Characteristics of stool will also be recorded for the three days prior to sampling using the Bristol criteria.

All food and drink intake will be recorded for the 7-day period prior to providing the first sample (baseline). Subjects will repeat this procedure at each sampling period. During the initial recording period, subjects will be asked to consume foods that represent their usual diet, with no more than a combined 4 fruit and vegetable servings each day, and be instructed to attempt to mimic the same diet during the 7 day periods each sampling period.

Diet records will be analyzed using nutrition software and the data will be used for analysis purposes as needed. Subjects will be encouraged to consume their usual diet throughout the study period.

Subjects will be weighed and total body composition determined using Dual-energy X-ray absorptiometry (DXA) for baseline subject characterization. Prior to the DXA scan a pregnancy test will be performed to confirm that the subject is not pregnant.

Subjects will be randomly assigned to supplement or the placebo capsules. The intervention will start between days 1 and 5 of the menstrual cycle to avoid confounding factors due to menstrual cycle hormone variation. The capsules are to be taken with a meal in the morning and in the evening with 3 capsules at each time, for a total of 6 capsules/day for a 20 week period. At the beginning of the 17th week, subjects consuming the supplement will be randomized with one group adding the "Complete" meal replacement component that will replace the first meal of the day and the second group following their normal diet.

Initial Laboratory Visit: screening visit During the initial visit to the laboratory, subjects will complete the informed consent form, health history, medication and dietary supplement usage and perceived stress questionnaires. Subjects' heart rate and blood pressure, height, weight, waist, and hip circumference will be measured. A pregnancy test will be performed to confirm that the subject is not pregnant. Body composition will be determined via DXA to determine body composition, as increased visceral fat is causative in obesity-induced inflammation. Upon completion of this screening visit, subjects will be scheduled for their initial testing visit.

Test Visit Procedures For each condition (supplement and placebo), subjects will report to the lab a total of three times. Subjects that continue on with the "Complete" meal-replacement phase of the study will report to the lab one additional time. Subjects will collect their stool during the 24 hours prior to reporting to the lab on each test occasion (or as close as possible to that time point). Subjects will report to the lab in a 10 hour fasted state, without having performed strenuous activity within the prior 48 hours. Subjects will have been instructed to obtain at least 7 hours of sleep during the night prior to testing. No supplement or placebo will be taken prior to blood collection, as described below.

Stool Collection Stool samples will be collected by subjects during the 24 hours immediately before reporting to the lab on each test occasion (or as close as possible to this time point). Subjects will be instructed to line the pail with the biohazard bag, complete a bowel movement in the bag, seal the bag with the zip tie, and place the bag in the insulated cooler bag with two freezer packs. The pail, biohazard bag, zip tie, insulated cooler and freezer packs will be provided by the investigator. Verbal and written instructions for collection, storage, and delivery of the stool samples will be available to each participant. Upon receipt by investigators, these samples will be stored at -70 degrees Celsius until processing. All sample handling will occur in the fume hood and universal precautions will be observed to minimize the risk of infection. Following publication of the study results, remaining stool samples will be disposed of properly as biohazard waste.

Blood Collection Blood samples (approximately 20 ml; 4 teaspoons) will be taken from subjects via venipuncture (by someone skilled in collecting blood). After the first blood draw, subjects will consume a cocktail of glucose, lactulose and mannitol. Another blood sample (3 ml) will be collected 90 minutes after ingestion of this cocktail. The purpose of consuming this cocktail and collecting a second blood sample is to determine the impact of the treatment on glucose tolerance and also its effect on intestinal permeability.

The collected blood samples will be processed and stored in multiple aliquots at -70 degrees Celsius until analyzed. Following publication of the study results, remaining blood samples will be disposed of properly as biohazard waste. Universal precautions will be observed to minimize the risk of infection or injury to either the subject or the phlebotomist. Potential risks for this procedure include soreness around the sampling site, bruising, and infection.

White Blood Cell Harvest White blood cells will be harvested from the collected whole blood using a density gradient (Ficoll) and stored in multiple aliquots at -70 degrees Celsius until analyzed. Following publication of the study results, remaining cell samples will be disposed of properly as biohazard waste. Universal precautions will be observed to minimize the risk of infection or contamination.

Dietary Intake and Records All subjects will be asked to consume their usual diet throughout the study period and be instructed to attempt to mimic the same diet during the 7 days prior to sampling. Subjects will record all food and drink consumed during the 7 days prior to each sampling day.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Critical care health care professional
* Premenopausal
* Overweight or obese (BMI: 25-40 kg/m2)
* Between the ages of 25-50

Exclusion Criteria:

* Smoking,including smokeless tobacco
* Chronic/excessive alcohol use
* Pregnant or lactating
* Recent surgery or illness
* Diabetes
* Heart disease
* Use of antibiotics

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2015-01; Primary Completion 2019-04-27 (Actual); Study Completion 2019-04-27 (Actual)

PRIMARY OUTCOMES:
Changes in intestinal microbiome composition induced by a fruit and vegetable supplement using 16S rRNA sequencing analysis | 1 year

SECONDARY OUTCOMES:
Changes in intestinal permeability by biochemical analysis | 1 year
Changes in systemic inflammatory molecules by cytokine analysis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marie van der Merwe, PhD, Principal Investigator — University of Memphis
Locations (1):
- The University of Memphis, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No